CLINICAL TRIAL: NCT06983223
Title: Oral Sucrosomial® Vitamin B12 in the Management of B12 Deficiency Among Metformin-Treated Type 2 Diabetes Patients: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Oral Sucrosomial® Vitamin B12 in the Management of B12 Deficiency Among Metformin-Treated Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LUMHS/REC/-733/09.05.2025
Record Dates: First submitted 2025-05-12; First posted 2025-05-21 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Vitamin B 12 Deficiency; Type 2 Diabetes Mellitus (T2DM)
Keywords: Metformin-Associated Vitamin B12 Deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled clinical trial. Participants will be randomly assigned in a 1:1 ratio to receive either Sucrosomial® B12 (1,000 mcg) or placebo once daily for 4 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be double-blind, meaning neither the participants, care providers, investigators, nor outcomes assessors will know the treatment allocation.
  Sucrosomial® B12 and placebo will be identical in appearance, packaging, and labeling to maintain blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sucrosomial® B12 Group (Experimental): Participants in this group will receive Sucrosomial® Vitamin B12 (1,000 mcg), administered as an orally dissolving powder, once daily for 3 weeks.
  Dosage Form: Orally dissolving powder (sachet) Administration Route: Oral
  Frequency: Once daily
  Duration: 3 weeks (21 days)
  Interventions: Dietary Supplement: Sucrosomial® Vitamin B12
- Placebo Group (Placebo Comparator): Participants in this group will receive a matching placebo (identical in appearance, packaging, and taste), administered as an orally dissolving powder, once daily for 3 weeks.
  Dosage Form: Orally dissolving powder (sachet)
  Administration Route: Oral
  Frequency: Once daily
  Duration: 3 weeks (21 days)
  Interventions: Other: Placebo (Oral)

INTERVENTIONS:
Dietary Supplement: Sucrosomial® Vitamin B12 — Sucrosomial® B12 is an advanced oral vitamin B12 supplement formulated with Sucrosomial® technology to enhance absorption. Participants in this group will receive 1,000 mcg of Sucrosomial® B12 (single sachet of orally dissolving powder) once daily for 3 weeks.
  Other Names: Oral Sucrosomial® Vitamin B12
  Arms: Sucrosomial® B12 Group
Other: Placebo (Oral) — Participants in the placebo group will receive an identical powder that matches the Sucrosomial® B12 in appearance, packaging, and administration. The placebo will be administered once daily for 3 weeks.
  Other Names: Matching Placebo
  Arms: Placebo Group

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the effectiveness of Sucrosomial® Vitamin B12 supplementation in the management of vitamin B12 deficiency among metformin-treated Type 2 Diabetes Mellitus (T2DM) patients. The study will compare the impact of daily Sucrosomial® B12 (1,000 mcg) versus placebo on serum vitamin B12 levels, Holo-Transcobalamin II (HoloTCII), and Transcobalamin I (TCI) levels over a 4-week period. Secondary outcomes include assessment of safety, tolerability, and glycemic control (HbA1c). Fifty participants will be randomly assigned to either the Sucrosomial® B12 or placebo group.

DETAILED DESCRIPTION:
Vitamin B12 deficiency is a common concern in Type 2 Diabetes Mellitus (T2DM) patients, especially those treated with metformin, which is known to interfere with B12 absorption. Early identification and effective management of B12 deficiency are critical to prevent neurological and hematological complications.

This study is designed as a randomized, double-blind, placebo-controlled clinical trial to assess the efficacy of Sucrosomial® Vitamin B12 (1,000 mcg daily) compared to placebo in improving vitamin B12 status among metformin-treated T2DM patients. The study will enroll 50 participants (25 in each group) who will receive either Sucrosomial® B12 or placebo for 4 weeks.

Primary Outcome:

Change in serum vitamin B12 levels from baseline to 3 weeks.

Secondary Outcomes:

Change in Holo-Transcobalamin II (HoloTCII) levels from baseline to 3 weeks.

Change in Transcobalamin I (TCI) levels from baseline to 3 weeks.

Safety and tolerability, assessed through adverse event monitoring.

Change in glycemic control (HbA1c) from baseline to 3 weeks.

The study will include assessments at Baseline, 24 hours, 7 days, 14 days, and 21 days. Blood samples will be collected at each time point to measure vitamin B12, HoloTCII, TCI, CBC, LFTs, and RFTs. The safety profile will be monitored throughout the study.

This study will provide essential data on the effectiveness of Sucrosomial® B12 in improving vitamin B12 status among metformin-treated T2DM patients, offering a potential non-invasive intervention for managing B12 deficiency in this population.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years.
* Diagnosed with Type 2 Diabetes Mellitus (T2DM).
* Currently on Metformin therapy for at least one year.
* Serum vitamin B12 levels below the laboratory reference range (indicating deficiency).
* Willing to provide written informed consent.
* Able to comply with study procedures and visit schedule.

Exclusion Criteria:

* Current or prior use of vitamin B12 supplements within the past 3 months.
* Diagnosis of pernicious anemia or other causes of vitamin B12 malabsorption (e.g., Crohn's disease, celiac disease).
* History of gastric surgery or small intestine resection.
* Use of medications known to interfere with vitamin B12 absorption (other than Metformin).
* Severe renal impairment (eGFR < 30 mL/min/1.73 m²) or end-stage renal disease.
* Severe hepatic impairment (ALT/AST > 3 times the upper limit of normal).
* Pregnant or breastfeeding women.
* Known hypersensitivity to vitamin B12 or any component of the study product.
* Participation in another clinical trial within the last 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Change in Serum Vitamin B12 Levels | Baseline, 24 hours, 7 days, 14 days, and 21 days.
  Assessment of change in serum vitamin B12 levels from baseline to 3 weeks.

SECONDARY OUTCOMES:
Change in Holo-Transcobalamin II (HoloTCII) Levels | Baseline, 24 hours, 7 days, 14 days, and 21 days.
  Change in Holo-Transcobalamin II (HoloTCII) Levels
Change in Transcobalamin I (TCI) Levels | Baseline, 24 hours, 7 days, 14 days, and 21 days.
  Assessment of Transcobalamin I (TCI) levels to evaluate the impact of Sucrosomial® B12 supplementation on vitamin B12 binding proteins. Blood samples will be collected at baseline, 24 hours, 7 days, 14 days, and 21 days.
Change in Gastric intrinsic factor levels | Baseline, 24 hours, 7 days, 14 days, and 21 days.
  Measurement of gastric intrinsic factor to assess the impact of Sucrosomial® B12 supplementation in metformin-treated Type 2 Diabetes patients.
Change in Holotranscobalamin (active B12) Levels | Baseline, 24 hours, 7 days, 14 days, and 21 days.
  Measurement of Holotranscobalamin to assess the impact of Sucrosomial® B12 supplementation in metformin-treated Type 2 Diabetes patients.
Incidence and Severity of Treatment-Emergent Adverse Events (Safety and Tolerability of Sucrosomial® B12) | Continuous monitoring throughout the 3-week intervention.
  Assessment of adverse events and side effects reported by participants during the 3-week intervention period. This includes the number of participants with one or more treatment-emergent adverse events (TEAEs), their severity (mild, moderate, severe), and the investigator-assessed relationship to the study product (Sucrosomial® B12).

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat University of Medical & Health Sciences (LUMHS), Jāmshoro, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Memon NM, Conti G, Brilli E, Tarantino G, Chaudhry MNA, Baloch A, Shafiq A, Mumtaz SU, Qaisar W, Iqtadar S, Abrar S, Kanwal A, Akhtar MH, Latif H, Rabbani F, Ujjan ID, Turroni S, Khan A. Comparative bioavailability study of supplemental oral Sucrosomial (R) vs. oral conventional vitamin B12 in enhancing circulatory B12 levels in healthy deficient adults: a multicentre, double-blind randomized clinical trial. Front Nutr. 2024 Nov 8;11:1493593. doi: 10.3389/fnut.2024.1493593. eCollection 2024. PMID 39582666
- [Background] Alhaji JH. Vitamin B12 Deficiency in Patients with Diabetes on Metformin: Arab Countries. Nutrients. 2022 May 13;14(10):2046. doi: 10.3390/nu14102046. PMID 35631186
- [Background] Sayedali E, Yalin AE, Yalin S. Association between metformin and vitamin B12 deficiency in patients with type 2 diabetes. World J Diabetes. 2023 May 15;14(5):585-593. doi: 10.4239/wjd.v14.i5.585. PMID 37273250
- [Background] Bell DSH. Metformin-induced vitamin B12 deficiency can cause or worsen distal symmetrical, autonomic and cardiac neuropathy in the patient with diabetes. Diabetes Obes Metab. 2022 Aug;24(8):1423-1428. doi: 10.1111/dom.14734. Epub 2022 May 20. PMID 35491956
- [Background] Gupta K, Jain A, Rohatgi A. An observational study of vitamin b12 levels and peripheral neuropathy profile in patients of diabetes mellitus on metformin therapy. Diabetes Metab Syndr. 2018 Jan-Mar;12(1):51-58. doi: 10.1016/j.dsx.2017.08.014. Epub 2017 Aug 25. PMID 28882470